CLINICAL TRIAL: NCT06484166
Title: Efficacy of Fullerene in Preventing Radiation Dermatitis in Patients With Head and Neck Cancer .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HX2024-134
Record Dates: First submitted 2024-06-24; First posted 2024-07-03 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis | interventions — triethanolamine; Biafine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trolamine (Biafine) (Active Comparator): Trolamine (Biafine; Genmedix Ltd, France) is cream packed in an opaque white bottle of 50g each, which is the same as the experimental group in appearance.
  Interventions: Drug: Trolamine (Biafine)
- Fullerene cream (Experimental): Fullerene cream is cream packed in an opaque white bottle of 50g each, which is the same as the control group in appearance.
  Interventions: Other: Fullerene cream

INTERVENTIONS:
Other: Fullerene cream — Patients are instructed to apply a thin layer of the Fullerene cream third a day, starting three days before radiotherapy(RT) and continue until two weeks after treatment. The application should include the whole treatment area. Patients are also advised to not apply the cream within four hours before the RT in order to avoid possible build-up effect. Patients are asked to keep the skin of the radiotherapy area dry and clean and not use other topical agents in the irradiated area.
  Arms: Fullerene cream
Drug: Trolamine (Biafine) — Patients are instructed to apply a thin layer of the Trolamine (Biafine) third a day, starting three days before radiotherapy(RT) and continue until two weeks after treatment. The application should include the whole treatment area. Patients are also advised to not apply the cream within four hours before the RT in order to avoid possible build-up effect. Patients are asked to keep the skin of the radiotherapy area dry and clean and not use other topical agents in the irradiated area.
  Arms: Trolamine (Biafine)

SUMMARY:
Radiotherapy always results in many complications such as radiation dermatitis, dry mouth, cranial nerve damage, and swallowing function. Among them, radiation dermatitis is confirmed to occur in the majority of tumor patients receiving radiotherapy, which not only affects the appearance but also causes the interruption of radiotherapy in severe cases.

At present, there is no standard treatment for radiation dermatitis. Trolamine is commonly prescribed at the beginning of radiotherapy for preventing acute radiation-induced skin toxicity in China. Fullerene cream is able to remove free radicals produced during radiotherapy, which may provide a new way and method for the prevention and treatment of radiation dermatitis. In addition, the product has obtained a safety assessment report from a third-party testing organization, proving that it has fully met the applied human body standards.

This clinical trial studies the effect of Fullerene cream in preventing radiation dermatitis in Head and Neck Cancer, compared with trolamine.

DETAILED DESCRIPTION:
Radiotherapy (RT) is an important treatment for head and neck malignant tumors and can be used alone or in combination with chemotherapy as radical or adjuvant therapy. Complications such as radiation dermatitis, dry mouth, cranial nerve damage, and poor swallowing function can occur in patients with head and neck cancer undergoing radiotherapy. Data from previous retrospective studies have shown that up to 90% of patients with head and neck tumors will develop radiation dermatitis after radiotherapy. Radiation dermatitis may cause the radiotherapy interrupted and treatment time prolonged, which will ultimately affect the treatment outcome and overall quality of life.

At present, there is no standard treatment for radiation dermatitis. Trolamine (Biafine; Genmedix Ltd, France) is an oil-in-water emulsion that can enhance skin healing by recruiting macrophages and modifying the concentrations of various immunomodulators. In China, Trolamine is commonly prescribed at the beginning of radiotherapy for preventing acute radiation-induced skin toxicity.

Fullerene is hollow molecules made entirely of carbon, with the ability to remove free radicals produced during radiotherapy. At the same time, Fullerene cream contains active ingredients such as ecdoine and sodium hyaluronate, which can effectively promote collagen production and speed up the repair of damaged skin. In addition, the product has obtained a safety assessment report from a third-party testing organization, proving that it has fully met the applied human body standards.

This clinical trial studies the effect of Fullerene cream in preventing radiation dermatitis in Head and Neck Cancer, compared with trolamine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients pathologically diagnosed with non-metastatic head and neck malignant tumors;
2. Patients considered candidates for high-dose RT either as primary treatment or as postoperative treatment after surgical resection and patients planned to receive concomitant boost fractionation or concurrent systemic chemotherapy.

Exclusion Criteria:

1. Eastern Cooperative Oncology Group performance status of >2;
2. Pre-existing skin rash, ulceration or open wound in the treatment area;
3. Known allergy to trolamine or fullerene;
4. Inflammatory or connective tissue disorder of the skin;
5. History of head and neck radiotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
The incidence of grade 2 or higher radiation dermatitis. | From the start of radiotherapy to 4 weeks after completion of radiotherapy.
  Patients are assessed weekly for radiation dermatitis by an experienced radiation oncology nurse according to the Radiation Therapy Oncology Group (RTOG) scale. The RTOG scale categorizes acute skin toxicity into grades 0-4, with the higher the grade the more severe the patient's acute radiation dermatitis. Grade 0 means no change over baseline. Grade 1 means follicular, faint, or dull erythema; epilation, dry desquamation, or decrease in sweating. Grade 2 means tender, bright erythema; patchy, moist desquamation or moderate edema. Grade 3 means confluent, moist desquamation other than skin folds; pitting edema. Grade 4 means ulceration, hemorrhage, necrosis.

SECONDARY OUTCOMES:
The time to onset of grade 2 or higher radiation dermatitis. | From the start of radiotherapy to 4 weeks after completion of radiotherapy.
  Time from the first day of radiotherapy to the first determination of grade 2 or higher radiation dermatitis.
The duration of grade 2 or higher radiation dermatitis. | From the start of radiotherapy to 4 weeks after completion of radiotherapy.
  The first determination of grade 2 or higher radiation dermatitis to the first instance of grade 1 or 0 radiation dermatitis, without a subsequent instance of grade 2 or higher radiation dermatitis. Patients without observed grade 2 or higher radiation dermatitis were assigned a duration of 0 days.
The maximum skin toxicity. | From the start of radiotherapy to 4 weeks after completion of radiotherapy.
  The maximum grade of RTOG skin toxicity between 0 and 4.
The Skindex-16 instrument. | From 1 week before radiotherapy to 4 weeks after completion of radiotherapy.
  The Skindex-16 is a commonly used tool to measure the effect of skin diseases on the QoL of patients. Skindex-16 consists of domain scores that assess how symptoms, emotions, and functioning from the skin issue affect the QOL of patients with acne. The overall score averages the 3 domain scores, all of which are normalized to a 0 to 100 scale, where 0 indicates that their skin condition has no impact on QOL and 100 represents maximal impact on QOL for the worse.
EORTC QLQ-C30. | From 1 week before radiotherapy to 4 weeks after completion of radiotherapy.
  The EORTC QLQ-C30 consists of five functional scales, nine symptom scales and one global quality of life (QoL) scale, and has been validated in an international setting.The questionnaire uses a four-point Likert scale to indicate the extent of problems experienced, ranging from 'not at all' to 'very much'. The answers for each domain are converted to a score ranging from 0 to 100；or functional scales, high scores represent a high level of QoL，and for symptom scales high scores indicate a poor QoL.
EORTC QLQ-H&N35 | From 1 week before radiotherapy to 4 weeks after completion of radiotherapy.
  The EORTC QLQ-H&N35 covers issues specific to HNC patients and includes 18 symptom scales; it has been validated in an international setting and is used extensively in HRQoL research. The questionnaire uses a four-point Likert scale to indicate the extent of problems experienced, ranging from 'not at all' to 'very much'. The answers for each domain are converted to a score ranging from 0 to 100；or functional scales, high scores represent a high level of QoL，and for symptom scales high scores indicate a poor QoL.
Adverse events. | From 1 week before radiotherapy to 4 weeks after completion of radiotherapy.
  Common Terminology Criteria for Adverse Events (CTCAE) 5.0 version.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No